CLINICAL TRIAL: NCT04790006
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Multiple Ascending Dose Phase Ib Study in Subjects With Type 2 Diabetes to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of TG103 Injection
Brief Title: A Study of TG103 in Subjects With Type 2 Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSA1803-CSP-003
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG103 (Experimental): TG103 will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Interventions: Drug: TG103
- Placebo (Placebo Comparator): Placebo will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TG103 — Administered SC
  Arms: TG103
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of multiple ascending doses of TG103 in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multicenter, dose-escalating study to characterize the safety (including the anti-drug antibodies(ADA)), tolerability pharmacokinetics (PK) and pharmacodynamic parameters（PD）of TG103. The study will consist of 3 periods: an approximately 2-week lead-in period, followed by a 12-week treatment period, and a 3-week safety follow-up period. Three dose groups (7.5mg, 15mg and 22.5mg) of subjects will be enrolled and dosed sequentially; 12

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who fully understand the test content and possible adverse reactions and voluntarily participate in the trial and sign the informed consent form;
* 2.Age: 18 to 75 years of age inclusive; no gender limitation;
* 3. Weight：body mass index (BMI) within the range of 18.5-35 kg/m2 (inclusive), BMI = weight (kg) / height 2 (m2);
* 4. Patients have diagnosed with type 2 diabetes ≤ 3 years according to the World Health Organization (WHO1999) classification; and not on medication or without a history of regular medication for more than 1 week in the 3 months prior to screening (subjects with a history of medication only include those with a history of oral medication and a history of short-term intensive insulin therapy (≤ 2 weeks));
* 5. 7.0% ≤ HbA1c ≤ 10.0%;
* 6. Subjects of childbearing potential must use reliable methods of contraception from the date of signing an informed consent to at least 3 months after the last dose;
* 7. The subject has the ability to communicate properly with the researcher and willing to fully comply with the research protocol.

Exclusion Criteria:

* 1. Fasting plasma glucose ≥13.9mmol/L or a history of severe hypoglycemia (blood sugar below 2.2mmol/L);
* 2. Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg during screening;
* 3. During the screening period, the white blood cell count fall outside the reference range by 10%, or hemoglobin<100g / L;
* 4. Have one or more positive tests in Hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti- Treponema pallidum-specific antibody;
* 5. Aspartate aminotransferase(AST) or Alanine aminotransferase (ALT) > 2.5x upper limit of normal (ULN), or triglyceride > 5.7mmol/L or eGFR<60 mL/（min*1.73 m2）during the screening period;
* 6. Hypercortisolism, polycystic ovary syndrome, abnormal thyroid function (those who need to be given medication or who have not reached clinical stability after treatment and whose medication still needs to be adjusted), etc. or other diseases that may affect blood glucose metabolism.
* 7. Have a personal or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia, or other genetic diseases that are susceptible to medullary cancer; personal or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia, or other genetic diseases that are susceptible to medullary cancer;
* 8. Acute complications of diabetes (including diabetic ketoacidosis, hyperosmolar nonketotic diabetic coma, lactic acidosis and hypoglycemia coma);
* 9. Proliferative diabetic retinopathy, foot ulcers/gangrene, and manifestations of peripheral neuropathy with obvious symptoms (e.g., gastroparesis, urinary retention, intestinal obstruction, urinary incontinence, and painful peripheral neuropathy);
* 10. Lost more than 400 ml of blood due to blood donation or other reasons within 3 months before the screening period;
* 11. During 3 months prior to screening through the entire study period, subjects used or plan to use drugs that may affect blood glucose metabolism or directly reduce gastrointestinal motility (e.g., anticholinergic drugs, antispasmodic, 5-HT3 antagonists, dopamine antagonists, and opioids), or oral and intramuscular injections of systemic corticosteroids, or inhalation or intranasal use of potent steroidal drugs with high systemic absorption; subjects regularly used thiazide diuretics within the 3 months prior to screening (Continuous medication > 1 week), or will use high doses of thiazide diuretics during the study period (hydrochlorothiazide>100 mg/d, chlorothiazide> 2 g/d, indapamide> 5 mg/d, chlorthalidone> 100 mg/d);
* 12. During the screening period, subjects with second degree or third degree atrioventricular block (except for subjects who use the pacemaker), long QT syndrome or prolonged QTc interval (male>450ms, female>470ms), or those with significant clinical symptoms of ischemic heart disease; or those with other heart diseases that are judged by the investigator to be unsuitable for entry into the study;
* 13. Any of the following cardiovascular and cerebrovascular events within half a year before screening: unstable angina pectoris requiring hospitalization, myocardial infarction, coronary artery bypass grafting, percutaneous coronary intervention (diagnostic angiography is allowed), moderate to severe congestive heart failure (NYHA grade III or IV), atrial or ventricular arrhythmia requiring hospitalization (such as atrial fibrillation and ventricular tachycardia). Subjects with pacemaker or defibrillator implantation, transient ischemic attack or cerebrovascular accident (e.g. stroke), or those with coronary artery bypass grafting or revascularization planned during the study period;
* 14. Have chronic or acute pancreatitis ( or have a history of chronic pancreatitis or acute pancreatitis) or severe gastrointestinal disease, such as confirmed reflux esophagitis or gallbladder disease, or any impact on gastric emptying (such as gastric bypass surgery, pyloric stenosis, except for appendectomy) or gastrointestinal diseases that may be aggravated by GLP-1 analogues; for patients with a history of gallbladder stones (gallstone removal or lithotripsy) and/or cholecystectomy, if there are no further sequelae, the entering of the study will be determined by researchers after assessing the risk;
* 15.Have a history of severe respiratory, blood system, and central nervous system (e.g. epilepsy) diseases; or have a history of malignant tumors or mental illnesses (such as depression, anxiety, etc.); or have other medical conditions that may endanger the safety of the subject and the investigator believes it is not suitable for inclusion;
* 16. Have had undergone major surgery within 3 months before screening, or had ongoing severe or acute infection within 4 weeks before screening;
* 17. Have a serious history of drug or food allergy, or may be allergic to the investigational product according to the judgment of the researcher;
* 18. Have taken prescription or over-the-counter medications for weight loss (e.g., orlistat, sibutramine, rimonabant, phenylpropanolamine, or chlorambucil) within 3 months prior to screening; or have undergone surgery that can cause weight instability; or have had a significant change in weight (>10% change);
* 19. Average alcohol intake is more than 21 units of alcohol (male)/14 units of alcohol (female) per week (1 unit ≈ 360mL beer, or 45mL spirits with 40% alcohol content, or 150mL wine) within the 3 months prior to screening;
* 20. Regularly consumption of caffeine is more than 600 mg of per day within the 3 months prior to screening (1 cup of coffee contains about 100 mg of caffeine, 1 cup of tea contains about 30 mg of caffeine, and 1 can of cola contains about 20 mg of caffeine);
* 21. Smoke more than 20 cigarettes per day within 3 months prior to screening;
* 22. Have skin abnormalities (such as: dermatitis) within a radius of 2cm of the administration site;
* 23.Participated in other clinical trial involving an investigational product within 3 months before the screening and the time of the last dose of the study drug is less than 3 months before the screening of this trial; or subjects withdrawn from the previous study due to an adverse event; or plan to participate other clinical trial during the study period;
* 24. Pregnant (blood pregnancy test positive in screening period) and lactating female;
* 25. Not suitable for this study in the researcher's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability assessed by incidence and severity of adverse events | up to 15 weeks
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Day1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78
  PK parameters after administration of of TG103
glycosylated hemoglobin (HbA1c) | Day15, 29, 43, 57,71, and 78,
  Pharmacodynamic (PD) parameters after administration of of TG103
The occurrence of TG103 anti-drug antibodies (ADA) | up to 15 weeks
  AD Aafter administration of of TG103
Peak Plasma Concentration (Cmax), | Day1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78
  PK parameters after administration of of TG103
Time to maximum plasma concentration (Tmax) | Day1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78
  PK parameters after administration of of TG103
Half time (t1/2), | Day1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78
  PK parameters after administration of of TG103
Apparent clearance (CL/F) | Day1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78
  PK parameters after administration of of TG103

CONTACTS AND LOCATIONS:
Overall Officials: Wenying Yang, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No